CLINICAL TRIAL: NCT05706467
Title: The Difference Between Non-invasive High-frequency Oscillatory Ventilation and Non-invasive Continuous Airway Pressure Ventilation in COVID-19 With Acute Hypoxemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Jianyi Niu, Principle investigator, Guangzhou Institute of Respiratory Disease
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYFYY-202301
Record Dates: First submitted 2023-01-28; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Pneumonia; Non-invasive Ventilation
Keywords: Noninvasive high frequency oscillatory ventilation; COVID-19 Pneumonia; acute hypoxic respiratory failure

STUDY DESIGN:
Intervention Model Description: Subjects who met the inclusion criteria received two kinds of non-invasive positive pressure ventilation treatment, namely, non-invasive continuous positive pressure ventilation and non-invasive high-frequency oscillatory ventilation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-invasive high-frequency oscillatory ventilation (Experimental): The day before the test, the patient was titrated with the oxygen concentration under non-invasive ventilation. The non-invasive continuous positive airway pressure ventilation was used, the pressure was set at 8cmH2O, and the oxygen concentration was titrated when the blood oxygen saturation was greater than 92% during non-invasive ventilation, and the oxygen concentration in the respiratory tube was constant after the test. In non-invasive high-frequency oscillatory ventilation mode, maintain the same positive airway pressure setting, and superimpose high-frequency oscillatory airflow with amplitude of 6cmH2O and oscillatory frequency of 10HZ.
  Interventions: Device: Non-invasive high-frequency oscillatory ventilation
- continuous positive airway pressure ventilation (Active Comparator): The patient was titrated with non-invasive ventilator-related parameters and oxygen uptake concentration the day before the test, and the parameter setting was maintained in the formal experiment.
  Interventions: Device: Non-invasive continuous positive airway pressure ventilation

INTERVENTIONS:
Device: Non-invasive high-frequency oscillatory ventilation — Non-invasive high-frequency oscillatory ventilation generates high-frequency pressure fluctuations in the airway caused by the opening and closing of a solenoid valve.
  Arms: non-invasive high-frequency oscillatory ventilation
Device: Non-invasive continuous positive airway pressure ventilation — Non-invasive positive airway pressure ventilation is carried out through non-invasive ventilator.
  Arms: continuous positive airway pressure ventilation

SUMMARY:
High frequency oscillatory ventilation (HFOV), as an ideal lung protection ventilation method, has been gradually applied to neonatal intensive care treatment, and is currently recommended as a rescue method for neonatal acute respiratory distress syndrome (ARDS) after failure of conventional mechanical ventilation. Although its ability to improve oxygenation and enhance carbon dioxide (CO2) clearance has been repeatedly demonstrated in laboratory studies, its impact on the clinical results of these patients is still uncertain. Noninvasive high-frequency oscillatory ventilation (nHFOV) combines the advantages of HFOV and non-invasive ventilation, and has become the current research focus in this field. It is recommended to use it after the failure of routine non-invasive ventilation treatment to avoid intubation. For the treatment of intubation, there is still a lack of large-scale clinical trials to systematically explore its efficacy. The gradual increase of clinical application of nHFOV has also enriched its application in the treatment of other diseases. At present, non-invasive high-frequency oscillatory ventilation has not been applied to the study of adult COVID-19 with acute hypoxemia, which will be the first study in this field.

ELIGIBILITY:
Inclusion Criteria:

1. After COVID-19 nucleic acid detection, imaging confirmed COVID-19;
2. Age ≥ 18 years old;
3. At the time of admission, the blood gas was acute hypoxic respiratory failure, the fraction of inhaled oxygen concentration (Fio2) was at least 0.40, but the blood oxygen saturation (Spo2) was 94% or lower;
4. Be able to follow the instructions of the researcher.

Exclusion Criteria:

1. Critically ill patients: cardiac and respiratory arrest, requiring tracheal intubation; Multiple organ failure (>2 organs);
2. Hemodynamic instability;
3. After extubation of invasive mechanical ventilation;
4. Patients who cannot wear a mask, such as maxillofacial or upper airway surgery;
5. Patients who may affect the treatment effect of NPPV, such as nasal obstruction or upper respiratory tract obstruction;
6. Obvious bullae, pneumothorax and pleural effusion;
7. It is accompanied by obvious other respiratory diseases, such as bronchiectasis and lung cancer;
8. Those who refuse to participate in this test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-10 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
ROX index | 30 minutes
  (SpO2/FiO2)/RR

SECONDARY OUTCOMES:
Asynchrony index | 30 minutes
  Asynchrony index is defined as the number of asynchrony events divided by the total respiratory rate computed as the sum of the number of ventilator cycles (triggered or not) and of wasted efforts: asynchrony Index (expressed in percentage) = number of asynchrony events/total respiratory rate (ventilator cycles +wasted efforts) × 100

CONTACTS AND LOCATIONS:
Overall Officials: Jianyi Niu, M.D., Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University. Guangdong, China